CLINICAL TRIAL: NCT05929508
Title: Improving Mobility and Function Following Transfemoral Amputation: A Novel Approach to Reverse Volumetric Muscle Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Lindsay Hannigan, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-0250
Record Dates: First submitted 2023-06-16; First posted 2023-07-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Amputation of Lower Extremity
MeSH Terms: interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic Preconditioning at High Pressure (Active Comparator): In this arm, the participant will receive ischemic preconditioning (a blood pressure cuff on the intact limb) inflated to 225mmHg for 5 minutes followed by 5 minutes of reperfusion on a cycle for a total of 50 minutes. This will be completed every other day for 7 session (14 days).
  Interventions: Other: Ischemic Preconditioning
- Ischemic Preconditioning at Low Pressure (Sham Comparator): In this arm, the participant will receive ischemic preconditioning (a blood pressure cuff on the intact limb) inflated to 25mmHg for 5 minutes followed by 5 minutes of reperfusion on a cycle for a total of 50 minutes. This will be completed every other day for 7 session (14 days).
  Interventions: Other: Ischemic Preconditioning

INTERVENTIONS:
Other: Ischemic Preconditioning — A blood pressure cuff will be placed on the thigh of the intact/sound limb to restrict blood flow to the lower extremity for 5 minutes and then deflated for 5 minutes to allow for normal blood flow on a cycle for 50 minutes (5 times).

SUMMARY:
The purpose of this study is to investigate the relationship between thigh strength and walking ability and assess if using a blood pressure cuff on the leg improves strength and walking performance.

DETAILED DESCRIPTION:
One in every 190 Americans is currently living with the loss of a limb. Following lower limb amputation (LLA), individuals have double the risk of knee and hip pain, a high prevalence of osteoarthritis in the intact limb with a prevalence ratio of 3.3 compared to those without amputation, and up to 90% experience severe back pain. The long-term consequences of LLA may be mitigated through regular use of prosthesis and physical activity, which would also increase the likelihood of returning to work and reintegration of Service Members (SMs) and younger Veterans.

Clinicians and researchers often focus on the prosthetic fit to improve outcomes, however just providing a prosthetic, even the most advanced prosthetic, is not enough to restore function. Interventions targeting physical capabilities to complement device intervention may be key to improving outcomes in individuals with LLA.

Along with increased orthopaedic risks, individuals with traumatic LLA also have an increased risk of cardiovascular events compared to the general population. SMs with traumatic unilateral transfemoral amputation have a 1.58 times greater risk of death from cardiovascular causes and their relative risk of aortic aneurysm is 5.1 times greater than Veterans without amputation. There is evidence to suggest that individuals with LLA have increased peripheral vascular resistance following amputation, leading to vasoconstriction and increased blood pressure. Reduced arterial function (i.e. increased arterial stiffness) is an important measure in those with LLA because it predicts mortality, heart failure, and cardiovascular events. In addition, improved arterial function improves perfusion to muscle and reduces fatigue during exertion. Therefore, strategies that reduce arterial stiffness and vascular resistance in individuals with LLA are important to improve mortality and quality of life for SMs and Veterans.

Therefore, we propose implementing ischemic preconditioning (IC) as a novel intervention to strengthen and hypertrophy leg muscles and increase arterial function for improving outcomes after amputation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* History of lower limb unilateral transfemoral amputation.
* At least two years post lower limb amputation
* Able to ambulate independently without the use of aids (i.e., walking cane).
* Able to walk at least 10 minutes continuously without stopping.
* Has a safe residuum with no open wounds on either the residual or intact limb.
* Has a prosthetic limb with materials that are sound and safe to withstand the mobility requirements of the study.

Exclusion Criteria:

* Younger than 18 years old.
* Inability to give informed consent.
* Neurological disorder that affects gait.
* Participants with significant metal (greater than one orthopaedic screw) in either the residual limb or the sound/intact limb
* Participants who begin taking medications or change dosage of medications that could affect gait, balance, and cardiovascular function during the course of the study.
* Currently pregnant (or intend to become pregnant while participating in study).
* History of any condition where fatiguing contractions or resisted leg contractions are contraindicated.
* Blood clots in the leg, or any condition in which compression of the thigh or transient ischemia is contraindicated (e.g. open wounds in the leg).
* History of uncontrolled hypertension.
* History of heart failure.
* Head injury within the previous 6 months.
* Seizure disorder.
* History of vascular disease.
* History of thrombosis.
* History of sickle cell trait.
* History of genetic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Strength | through study completion, an average of 6 weeks
  Comparing leg strength before and after intervention
Gait | through study completion, an average of 6 weeks
  Comparing leg strength before and after intervention
Metabolics | through study completion, an average of 6 weeks
  Comparing leg strength before and after intervention
Daily Steps/Activity | through study completion, an average of 6 weeks
  Comparing leg strength before and after intervention
Arterial Stiffness | through study completion, an average of 6 weeks
  Comparing leg strength before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Slater, Principal Investigator — University of Illinois at Chicago
Locations (1):
- UIC Physical Therapy Faculty Practice, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No